CLINICAL TRIAL: NCT00468637
Title: Association of Multiple CardiOvascular Risk Factors and Erectile Function Across Europe
Acronym: AMORE-Eur
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Saarland (Other)
Collaborators: Pfizer (Industry)
Responsible Party: Dr. Magnus Baumhäkel, Department of Cardiology, University Hospital of the Saarland
Other Study IDs: 133/04
Record Dates: First submitted 2007-05-02; First posted 2007-05-03 (Estimated); Last update posted 2009-02-16 (Estimated); Status verified 2009-02

CONDITIONS: Cardiovascular High-Risk; Chronic Heart Failure
Keywords: heart failure; cardiovascular high risk; erectile dysfunction; cardiovascular disease
MeSH Terms: conditions — Heart Failure; Erectile Dysfunction; Cardiovascular Diseases

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of the study is to evaluate the influence of cardiovascular risk factors, heart failure and cardiovascular drug therapy on erectile function in cardiovascular high-risk patients.

DETAILED DESCRIPTION:
Association of cardiovascular risk factors and ED is likely due to an impairment of endothelial function resulting in a decreased activity of endothelial NO-synthase, which plays a major role in physiology of erection. Heart failure is also known to further contribute to endothelial dysfunction and hence, this could lead to erectile dysfunction.

Study Objectives

1. Evaluation of the influence of cardiovascular risk factors and concomitant medication on erectile function in cardiovascular high-risk patients.
2. Evaluation of the role of heart failure on prevalence and severity of erectile dysfunction in men.
3. Long-term effects of cardiovascular drug therapy and cardiovascular diseases on erectile function.

Study Design Male patients across Europe with cardiovascular diseases (CHD, PAD and heart failure) will be evaluated with a standardized questionnaire. Grade of erectile dysfunction will be assessed using an ED-score, generated from two different questionnaires.

1. IIEF-5 - (International Index of Erectile Function)
2. KEED - (Cologne Evaluation of Erectile Dysfunction)

Primary Endpoint The primary endpoint is the sum score of the ED rating scale of the KEED (Kölner Erhebungsbogen zur Erektilen Dysfunktion, see Appendix 1). Erectile dysfunction is defined as reaching more than 17 points in the sum score.

Secondary Endpoint The first secondary endpoint is the frequency of sexual activity and sexual desire. Another secondary endpoint contains satisfaction with sex life and general well-being. Men are defined as dissatisfied by answering "mixed" or "worse".

Follow-Up: after 1 year, after 2 years.

ELIGIBILITY:
Inclusion Criteria:

* Male patients with two or more cardiovascular risk factors or
* Male patients with a manifestation of atherosclerosis or
* Male patients with an ischemic or dilated cardiomyopathy
* Written informed consent

Exclusion Criteria:

* Impairment of hormonal status
* Refusal of written informed consent
* Inability to complete the questionnaires

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: primary care clinic, outpatient department, general practitioner
Sampling Method: Non-Probability Sample
Enrollment: 1200 (Estimated)
Dates: Start 2007-05; Study Completion 2011-09 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Böhm, MD, Principal Investigator — Department of Cardiology, University Hospital of the Saarland; Magnus Baumhäkel, MD, Principal Investigator — Department of Cardiology, University Hospital of the Saarland
Locations (4):
- Germany (2):
  - Department of Cardiology, University Hospital of the Saarland, Homburg, Saarland
  - Gemeinschaftspraxis & Ambulante Tagesklinik, Merzig-Schwemlingen, Saarland
- Section on Cardiovascular Diseases, Department of Experimental and Applied Medicine, University of Brescia, Brescia, Italy
- Department of Cardiology, 4th Military Clinical Hospital, Wroclaw, Poland

REFERENCES:
- [Background] Rosen RC, Cappelleri JC, Smith MD, Lipsky J, Pena BM. Development and evaluation of an abridged, 5-item version of the International Index of Erectile Function (IIEF-5) as a diagnostic tool for erectile dysfunction. Int J Impot Res. 1999 Dec;11(6):319-26. doi: 10.1038/sj.ijir.3900472. PMID 10637462
- [Background] Braun M, Wassmer G, Klotz T, Reifenrath B, Mathers M, Engelmann U. Epidemiology of erectile dysfunction: results of the 'Cologne Male Survey'. Int J Impot Res. 2000 Dec;12(6):305-11. doi: 10.1038/sj.ijir.3900622. PMID 11416833
- [Background] Petrone L, Mannucci E, Corona G, Bartolini M, Forti G, Giommi R, Maggi M. Structured interview on erectile dysfunction (SIEDY): a new, multidimensional instrument for quantification of pathogenetic issues on erectile dysfunction. Int J Impot Res. 2003 Jun;15(3):210-20. doi: 10.1038/sj.ijir.3901006. PMID 12904808